CLINICAL TRIAL: NCT01139294
Title: Phase IV Randomized Study of Hylenex or Standard IV Hydration in the Pediatric Population With Moderate Dehydration
Brief Title: Descriptive Study of Cardiac Output During Rehydration With Recombinant Human Hyaluronidase in Pediatrics
Acronym: Hylenex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Thomas Abramo, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 091087; Clinical Trial (Other Grant/Funding Number: Baxter)
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Dehydration; Cardiac Output; Pediatrics
Keywords: cardiac output; dehydration; pediatrics
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard IV therapy (No Intervention): control arm of the study
- Hylenex (Experimental): 1ml subcutaneous with initiation of intravenous fluids then every 24 hours with a maximum dose of 3 injections in 72 hours
  Interventions: Drug: Hylenex

INTERVENTIONS:
Drug: Hylenex — 1ml subcutaneous with initiation of intravenous fluids then every 24 hrs with a maximum dose of 3 injections in 72 hours
  Other Names: hyaluronidase human injection
  Arms: Hylenex

SUMMARY:
The purpose of this study is to non-invasively study the reflective changes in cardiac output as response to fluid therapy in the pediatric moderate hypovolemia/dehydrated pediatric patients using sub-q rehydration using Hylenex augmented subcutaneous infusion of fluids and electrolytes compared to intravenous methods.

DETAILED DESCRIPTION:
This is an open-labeled, single-center Phase IV clinical trial. The study will consist of patients with moderate hypovolemia/dehydration requiring parenteral rehydration. It is expected that this study will describe the onset or change in cardiac output using Hylenex augmented subcutaneous rehydration from ages 2 months up to 3 years and at a flow rate satisfying clinical needs, especially in reference to changes in cardiac output observed in standard intravenous rehydration.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to the Emergency Department (ED) with moderate dehydration (gorelick dehydration classification : presence of 3-6 moderate signs and symptoms) requiring parenteral rehydration.
* Patient has not successfully received oral or IV fluids immediately prior to enrollment
* patient's legally authorized representative has signed the informed consent and is willing for the patient to receive Hylenex augmented sub-q rehydration

Exclusion Criteria:

* patient in shock or a life-threatening situation
* immunocompromised, history of abscess or cellulitis, abscess &/or cellulitis caused by Methicillin-resistant Staphylococcus aureus (MRSA), family history of abscess or cellulitis
* requires IV therapy for another indication
* has an indwelling catheter
* has already received rehydration therapy by IV route within the last 48 hours or substantial oral fluid in the immediate time period of enrollment
* has a condition precluding sub-q injection or infusion site evaluation in the upper middle back area or at another elected site of infusion
* has a reason for hospital admission or extended ED stay other than dehydration
* has an known hypersensitivity to hyaluronidase or another ingredient in the formulation of Hylenex
* has a know hyponatremia < 130 milliequivalents per liter (mEq/L) or hypernatremia >155 mEq/L
* has a know hypokalemia <3.0 mEq/L
* has a medical condition likely to interfere with the patients ability to fully complete the study protocol or the ability to have the protocol-specified assessments
* has a medical history, screening physical exam finding or historical clinical lab result that in the opinion of the investigator would preclude the patients safe participation in the is study or which might adversely effect the interpretation of the study results
* patient participated in a study of any investigational drug or device within 230 days prior to enrollment in this study

Ages: 2 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Abramo, MD, Principal Investigator — Monroe Carell Jr. Children's Hospital at Vanderbilt
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants were enrolled into the study per the final report to the Institutional Review Board. Actual study data was lost, so arm assignments are unknown.
Groups:
- Standard of Care IV Therapy: control arm of the study
- Hylenex: 1ml sub-q with initiation of IVF's then every 24 hrs with a max dose of 3 inj. in 72 hours
  Hylenex: 1ml sub-q with initiation of IVF's then every 24 hrs with a max dose of 3 inj. in 72 hours
Period: Overall Study
Arm/Group | Standard of Care IV Therapy | Hylenex
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No baseline data available. Study data was lost. Data was left behind when PI left institution in 2013. Unable to find anyone with knowledge of data location.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care IV Therapy | Hylenex | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Output Trends
Description: Describe the cardiac output trends measured in liters per minute (onset and changes in slope over time) by noninvasively monitoring methods in pediatric patients being rehydrated by Hylenex augmented subcutaneous rehydration or routine IV rehydration
Time Frame: Measurements and data are recorded only while patient is receiving care in the Emergency Department (ED). A f/u call is made on day 3 and/or day 7 post enrollment into the study.
Population: No outcome measure data available. Study data was lost. Data was left behind when PI left institution in 2013. Unable to find anyone with knowledge of data location.
Arm/Group | Standard of Care IV Therapy | Hylenex
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Gorelick Assessment
Description: Gorelick assessment of hydration status at baseline, and at the end of sub-q or IV hydration treatment or at discharge from the emergency dept.
  * volume of fluid infuse over time
  * time to discharge from ED to home or transfer into the hospital
  * discharge diagnosis from ED
  * duration of any supplemental hospitalization for supplemental hydration
  * time to first urine output observed
  * requirement for rescue therapy and nature of the rescue therapy
  * incidence of readmission to hospital/ED
  * global assessment of overall satisfaction with rehydration therapy by parents and caregiver
Time Frame: Measurements and data are recorded only while patient is receiving care in the ED. A f/u call is made on day 3 and/or day 7 post enrollment into the study.
Population: No outcome measure data available. Study data was lost.Data was left behind when PI left institution in 2013. Unable to find anyone with knowledge of data location.
Arm/Group | Standard of Care IV Therapy | Hylenex
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No adverse event data available. Study data was lost. Data was left behind when PI left institution in 2013. Unable to find anyone with knowledge of data location.
Arm/Group | Standard of Care IV Therapy | Hylenex
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study data was lost.Data was left behind when PI left institution in 2013. Unable to find anyone with knowledge of data location.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes